CLINICAL TRIAL: NCT01919762
Title: Detecting Infections Rapidly and Easily for Bacteremia Trial (DIREBT)-Part I (Prospective Collection and Freezing of Whole Blood Specimens)
Brief Title: Detecting Infections Rapidly and Easily for Bacteremia Trial (DIREBT)
Acronym: DIREBT
Status: Completed | Type: Observational
Sponsor: T2 Biosystems (Industry)
Responsible Party: Sponsor
Other Study IDs: PRO-00191
Record Dates: First submitted 2013-08-07; First posted 2013-08-09 (Estimated); Last update posted 2015-09-28 (Estimated); Status verified 2015-09

CONDITIONS: Bacteremia
Keywords: Bacteremia; Sepsis; Acinetobacter baumannii; Staphylococcus aureus; Klebsiella pneumonia; Pseudomonas aeruginosa; Enterococcus faecalis; Magnetic Relaxation Detection; Nuclear Magnetic Resonance Detection; Blood culture
MeSH Terms: conditions — Bacteremia; Sepsis; Staphylococcal Infections; Pseudomonas Infections

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood specimens, in addition to bacterial isoaltes
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Bacteremia Positive Patients: Symptomatic adult patients, confirmed via diagnostic blood culture and species identification followed by subsequent second blood culture results and species identification that are positive for each of the following species of bacteria (Target 6 Species).
  * Acinetobacter baumannii
  * Staphylococcus aureus
  * Klebsiella pneumonia
  * Pseudomonas aeruginosa
  * Enterococcus faecalis
  * Enterococcus faecium
- Bacteremia Negative Patients: Adult patients confirmed via diagnostic blood culture and species identification and subsequent second blood culture and species identification as being negative for the Target 6 species

SUMMARY:
To assure the uniform collection, handling, storage and transport of patient whole blood specimens and associated information to support validation of the T2 Bacteremia Assay.

DETAILED DESCRIPTION:
This protocol is intended for use by external sites collecting clinical research specimens for T2 Biosystems' use in developing the T2Bacterial Assay. Specimens and information on patients' medical history, blood properties, medications, and blood culture history/results are required from the T2Bacterial Assay's target patient population (i.e., candidates for blood culture). Ideally, clinical specimens for use in developing the T2Bacterial Assay will be collected from negative blood culture, positive non-bacteria blood culture and positive bacteria blood culture patients.

ELIGIBILITY:
Inclusion Criteria:

* Subject or subject's authorized representative must be able to understand, read and sign the study specific informed consent form after the nature of the study has been fully explained to them.
* Males and females 18 - 95 years of age.

For Group A,

* Subject is confirmed to have bacteremia (gram negative rods, gram negative coccobacillus, and/or gram positive cocci) as evidenced by a positive diagnostic blood culture
* Subsequent species identification identifies the presence of one of the following 6 species of bacteria:
* Acinetobacter baumannii
* Staphylococcus aureus
* Klebsiella pneumonia
* Pseudomonas aeruginosa
* Enterococcus faecalis
* Enterococcus faecium

For Group B,

* Males and females 18 - 95 years of age.
* Subject is confirmed to not have bacteremia from the 6 bacteria species targeted by this study, as evidenced by diagnostic blood culture and subsequent species identification.

Exclusion Criteria:

* Use of any novel (i.e. not commercially available) drug compound within 30 days prior to the collection of T2 blood specimens.
* Subject has other co-morbid condition(s) that, in the opinion of the Investigator, could limit the subject's ability to participate in the study or impact the scientific integrity of the study.
* Subject has had an anti-bacterial drug administered through the same port or central line as is used to collect the clinical research specimens. A line draw cannot be used to obtain a study sample if an antibacterial agent was administered intravenously within the last 72 hours, unless the site can specifically document that a different line was used to administer the anti-bacterial agent.

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with blood culture results are eligible to participate
Sampling Method: Non-Probability Sample
Enrollment: 156 (Actual)
Dates: Start 2013-08; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Number of bacteremia positive patients | 3-5 days post blood culture
  Number of bacteria positive patients based on concordant, sequential blood culture results and a positive T2 signal

SECONDARY OUTCOMES:
Number of bacteremia negative patients | 3-5 Days post blood culture
  Number of negative bacteremia samples based on concordant, sequential blood culture results and a negative T2 signal

CONTACTS AND LOCATIONS:
Locations (1):
- Cooper Medical School, Camden, New Jersey, United States